In vivo study for the evaluation of the efficacy of an adjunct mouthwash in hygiene, wound healing, analgesia, and functional recovery following trauma or dental procedures in gingival tissue.

**Protocol ID:** 23-003-01

**Date:** 14Dec2023

## **Study synopsis**

The study was aimed to assess the efficacy of a cosmetic product in improving oral mucosa healing after dental intervention. In order to reach this goal a randomized, placebo controlled, blind, single centre study was carried out on 94 (100 enrolled) healthy female and male subjects more than 18 years old, enrolled according to the specific inclusion and non-inclusion criteria. The subjects had a dental procedure on oral mucosa tissue and used the mouthwash or placebo (according to the randomization list) for 15 days following the procedure. Efficacy evaluations were performed at baseline (T0), after 7 (T7) and 15 days (T15) of product use by means of the post procedure would aspect assessment grading on Likert scale, as well as the pain evaluation on the 0 to 10 scale. The study was approved by an independent ethics committee, and no protocol amendments were done after the approval.